CLINICAL TRIAL: NCT06991881
Title: Eosinophilic Esophagitis: Towards Improved Management
Acronym: EoStim
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Helse-Bergen HF (Other)
Responsible Party: Principal Investigator, Ketil Størdal, Dr, Oslo University Hospital
Other Study IDs: 201046
Record Dates: First submitted 2025-02-17; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Months
Biospecimen Retention: Samples With DNA — Blood samples (EDTA), serum samples, oesophageal biopsies and brushes, stool samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Biobank sampling for new biomarkers — Using biopsies as the gold standard, the project aims towards validating non-invasive biomarkers as specified previously against biopsies.

SUMMARY:
The current project aims to improve the care for children and adolescents with eosinophilic esophagitis in a collaborative effort involving pediatric units at Oslo Unversity Hospital and Helse Bergen, Norway. Existing and new non-invasive biomarkers will be explored systematically, aiming to reduce the number of endoscopies and time on restricted diet.

DETAILED DESCRIPTION:
The overall aim of the current proposal is to improve the care for children and adolescents with EoE and reduce the need for complex elimination diets and repeated endoscopies.

Our objectives are to determine whether

1. at diagnosis the following are predictive for response to food elimination:

   1. history of atopy, symptoms after food intake
   2. eosinophil counts in biopsies and peripheral blood
   3. total IgE, specific IgE, eosinophilic granula proteins, eosinophil progenitor cells in blood
   4. key cytokines (Eotaxin-3, IL-5, IL-13)
   5. eosinophil derived neurotoxin/EDN in oesophageal aspirates, blood samples and feces
   6. circulating microRNAs
2. at follow-up biomarkers collected by non-invasive methods can predict endoscopic and histologic healing

   1. eosinophil counts in esophageal brushes and peripheral blood
   2. total IgE, specific IgE, eosinophilic granula protein, eosinophil progenitor cells
   3. circulating cytokines like eotaxin-3, IL-5, IL-13
   4. eosinophil derived neurotoxin/EDN in esophageal brushes, blood samples and feces
   5. circulating microRNAs

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of eosinophilic esophagitis
* suspected but not yet confirmed eosinophilic esophagitis

Exclusion Criteria:

* chronic severe conditions that preclude general anaestesia
* lack of consent

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with newly diagnosed or previously confirmed eosinophilic esophagitis.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Active eosinophilic esophagitis (>15 eosinophils per high-power field) | 12 months
  The eosinophil counts in a biopsy is used to classify active vs non-active eosinophilic esophagitis, and biomarkers are analysed using biopsy the gold standard to classify active vs inactive disease.

CONTACTS AND LOCATIONS:
Overall Officials: Ketil Størdal, PhD, Principal Investigator — University of Oslo
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Bergen
  - OsloUH, Oslo

IPD SHARING:
Plan to Share IPD: No
Not planned due to confidentiality